CLINICAL TRIAL: NCT03566160
Title: Pilot Study for Evaluation of Cryobiopsy and Correlation With Standard Forceps Biopsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-P000734
Record Dates: First submitted 2018-05-25; First posted 2018-06-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Gastrointestinal Disease
Keywords: Biopsy; EGD; Endoscopy; Cryobiopsy; OCT
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cryobiopsy probe as a tool for biopsy (Experimental): Cryobiopsy probe, administered to study participants.Testing the efficacy of a novel cryobiopsy probe in acquiring tissue samples.
  Interventions: Device: Cryobiopsy probe, administered to study participants

INTERVENTIONS:
Device: Cryobiopsy probe, administered to study participants — Cryobiopsy probe as a tool for gastrointestinal biopsy

SUMMARY:
Environmental enteric dysfunction (EED) is a poorly understood condition characterized by intestinal inflammation and loss of barrier function that is prevalent in regions of the world with inadequate sanitation and hygiene. EED is a major driver of malnourishment, poor neurological development, stunting, oral vaccine failure, and infection, affecting 25% of all children globally and causing over a million deaths each year.

Progress towards understanding EED and developing effective interventions has been hampered by an inability to evaluate the intestinal mucosa of populations in impoverished regions of the world where this condition is endemic. In order to prevent the deleterious and permanent sequelae of the disease, there is a need for effective diagnosis and intervention to be implemented in EED patients before the age of 2. Currently, the only means for directly evaluating the intestine is endoscopy with mucosal biopsy. Unfortunately, endoscopy is untenable for the study of EED because of limited resources and the high cost. As a result, there is a clear, unmet need for a less invasive tool that can be used in low-and-middle-income-countries (LMICs) to evaluate the intestine in population with EED.

This work is supported by a grant from The Bill and Melinda Gates Foundation (BMGF). The overall goal is to provide a minimally invasive means of obtaining detailed infantile intestinal tissue information that is needed for the development of effective EED interventions. Obtaining biopsies will play a critical role in gathering the detailed intestinal tissue information.

The purpose of this study is to explore the feasibility of utilizing a cryobiopsy probe to obtain biopsies in adults.

DETAILED DESCRIPTION:
This study will test the capacity of a gastrointestinal tract cryobiopsy probe that Tearney Lab investigators have designed to obtain biopsies from the upper GI tract.

A total of twenty (20) participants, adults 18 years of age and older, scheduled for elective esophagogastroduodenoscopy with biopsy will be enrolled in this study.

A maximum of 3 cryobiopsies per subject will be collected. After each cryobiopsy is complete, the endoscopist will then take 1 standard forceps biopsy from the area adjacent to where cryobiopsy was performed. A maximum of 3 standard forceps biopsies for research purposes only will be taken. Biopsy collection will be performed at the discretion of the endoscopist. The standard forceps biopsy sites will also be monitored directly throughout the entire experimental procedure. The total experimental procedure time will not exceed 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an elective esophagogastroduodenoscopy with biopsy.
* 18 years of age or older.
* Able to provide informed consent.

Exclusion Criteria:

* According to standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Cryobiopsy probe | 3 years
  Evaluation of Cryobiopsy probe in obtaining tissue samples over .5mm

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No